CLINICAL TRIAL: NCT04265144
Title: Cohort of Patients With Systemic Sclerosis and Associated Biological Collection Within the Framework of the RESO Reference Centre for Rare Systemic Autoimmune Diseases
Brief Title: Cohort of Patients With Systemic Sclerosis Within the Framework of the RESO Reference Centre
Acronym: SCLERESO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2019/42
Record Dates: First submitted 2020-02-05; First posted 2020-02-11 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Scleroderma; Systemic Sclerosis
Keywords: Cohort study; systemic sclerosis; prognosis
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic | interventions — Blood Specimen Collection; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- subjects SSc diagnosed (Experimental): Patient with systemic scleroderma according to the American College of Rheumatology (ACR) / EULAR 2013 criteria
  Interventions: Biological: Blood samples; Other: Biopsy; Other: Bronchoalveolar samples

INTERVENTIONS:
Biological: Blood samples — 62 ml whole blood for Peripheral blood mononuclear cell (PBMC) and monocytes isolation
Other: Biopsy — Skin biopsies only for volunteers among patients
Other: Bronchoalveolar samples — 50 ml of bronchoalveolar samples if pulmonary flare requires this type of exploration only for volunteers among patients
Other: Biopsy — Digestives biopsies if requires this type of exploration in the standard of care only for volunteers among patients

SUMMARY:
Systemic sclerosis (SSc) is a rare form of connective tissue disease characterized by vascular involvement and the intensity of fibrosis. The lack of available treatment is largely due to the very fragmented understanding of the pathophysiology of SSc. However, one of the keys to conducting quality research on this disease remains the development of well-documented patient cohorts with reliable biological samples. The main objective of this cohort is to study the natural progression of SSc in a cohort of patients followed over 5 years.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a rare form of connective tissue disease characterized by vascular involvement and the intensity of fibrosis. Its prevalence and incidence are difficult to assess, however, in France, a population survey conducted in Seine-St-Denis calculated a prevalence of 161 cases per million inhabitants.

The pathophysiology of SSc, the exact etiology of which remains unknown, involves an interaction between genetic and environmental factors. Its evolution can impact the aesthetic, functional and even vital prognosis of the affected patient.Within the analysis of SSc pathophysiology, a " very early systemic sclerosis " form of disease has been defined according to the presence of Raynaud's phenomenon and auto-antibodies in blood sample (ACAN positivity (≥1/160) with anti-Scl70, anti-centromere or anti-ARNPolIII specificity).

At present, no treatment to control this disease is available. The lack of available treatment is largely due to the very fragmented understanding of the pathophysiology of SSc. However, one of the keys to research remains the development of well-documented patient cohorts with quality biological samples. The investigators had the opportunity to start a major work on this plan with the VISS study (Vasculopathy and Inflammation in Systemic Scleroderma study) in 2012 as part of a project promoted by the University Hospital of Bordeaux (NCT02562079). This project has paved the way for many local, national and international collaborations. It has made it possible to structure and federate various partners of the Bordeaux University Hospital around translational research on SSc.

The investigators wish to continue our research and collaborations by further strengthening our expertise in the collection of rare and valuable biological samples for this disease.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Patient with systemic scleroderma according to the ACR/EULAR 2013 criteria, or with a " very early systemic sclerosis " defined by the presence of Raynaud's phenomenon and auto-antibodies in blood sample (ACAN positivity (≥1/160) with anti-Scl70, anti-centromere or anti-ARNPolIII specificity).
* Person affiliated or benefiting from a social security scheme.
* Free, informed and written consent signed by the participant and the investigator (no later than the day of inclusion and prior to any review required by the research)

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Patient under guardianship, curatorship or any other legal protection regime

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-06-08 (Actual); Primary Completion 2034-06 (Estimated); Study Completion 2034-06 (Estimated)

PRIMARY OUTCOMES:
Change of the main clinical characteristics of scleroderma patients | At baseline (Day 0) and 60 months after baseline
  Worsening of the SSc according to the onset of a renal crisis (according to arterial hypertension > 150/85 mm Hg ), a pulmonary arterial hypertension (identified with a right heart catheterization), or an interstitial lung disease (identified with a chest CT-scan).

SECONDARY OUTCOMES:
Proportion of pulmonary arterial hypertension diagnosis in SSc patients | At baseline (Day 0) and 60 months after baseline
Proportion of interstitial lung disease diagnosis in SSc patients | At baseline (Day 0) and 60 months after baseline
Proportion of renal crisis diagnosis in SSc patients | At baseline (Day 0) and 60 months after baseline
Mean of Rodnan score for the evaluation of disease activity for SSc patients, with higher values mean higher disease activity. | At baseline (Day 0) and 60 months after baseline
  (Min value: 0 - Max value: 51)
Mean of Diffusing capacity (DLCO) for the evaluation of disease activity for SSc patients | At baseline (Day 0) and 60 months after baseline
Mean of Forced vital capacity (FVC) for the evaluation of disease activity for SSc patients | At baseline (Day 0) and 60 months after baseline
Proportion of therapeutic strategies set up for SSc patients | At baseline (Day 0) and 60 months after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Elise TRUCHETET, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux - service de rhumatologie, Bordeaux, France